CLINICAL TRIAL: NCT03026400
Title: Sub vs Trans-umbilical Incision: A Patient's Satisfaction-centered Randomised Trial
Brief Title: Sub vs Trans-umbilical Incision: A Patient's Satisfaction-centered Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-688
Record Dates: First submitted 2017-01-06; First posted 2017-01-20 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Patient Satisfaction; Surgical Wound; Incision; General Surgery
MeSH Terms: conditions — Patient Satisfaction; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subumbilical incision (Other): The subumbilical incision was standardised. A curvilinear horizontal incision was performed to be able to reach the base of the umbilicus. The aponeurosis was incised with a scalpel and the peritoneal layer was open with a Kelly clamp. The incision was completed with the Hasson technique and a X-stitch was used for closure.
  Interventions: Procedure: Subumbilical incision
- Transumbilical incision (Other): The transumbilical incision was also standardised, inverting the umbilicus with graspers, then incising vertically the skin to reach the umbilical physiological hernia to enlarge it. The incision was also completed with the Hasson technique and a X-stitch was used for closure.
  Interventions: Procedure: Transumbilical incision

INTERVENTIONS:
Procedure: Transumbilical incision — While both types of incision were considered equal regarding the potential clinical outcome, the investigators considered the transumbilical incision to be the ''intervention'' and the subumbilical incision to be the ''standard care comparator'' since the transumbilical incision take a few more minutes to be completed.
  Arms: Transumbilical incision
Procedure: Subumbilical incision — Considered here as the ''control'' intervention.
  Arms: Subumbilical incision

SUMMARY:
While some studies have suggested that subumbilical and transumbilical incisions have a similar clinical efficiency and safety, no study has yet evaluated their respective impact on patient's postoperative aesthetic satisfaction.

The objective of this randomised trial is to compare patient's postoperative aesthetic satisfaction depending on the type of incision which is performed during surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years old having a planned laparoscopic surgery with an umbilical first trocar at CHUS were included.

Exclusion Criteria:

* Patients with a BMI > 40 or that had previous abdominal surgeries involving the umbilicus were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in postoperative patient's aesthetic satisfaction | 6 months
  An inverted 10 points Wong-Baker facial grimace-type scale was used to assess patient's satisfaction. Although the french version of our questionnaire was not validated, the concept behind Wong-Baker facial scale have been in various studies. In the case of this study, a 10 point score was associated with the highest possible satisfaction regarding the aesthetic appearance of the umbilicus.
  Patient's aesthetic satisfaction regarding the umbilicus was recorded preoperatively (right before the surgery), 1 month post-op and 6 months post-op. The change in postoperative patient's aesthetic satisfaction was assessed between pre-op vs 1 month post-op, pre-op vs 6 months post-op and 1 month vs 6 months post-op.

SECONDARY OUTCOMES:
Level of patient's awareness regarding the aesthetic appearance of the umbilicus | Pre-operative
  YES/NO (no meaning that the patient gives little to no importance to the aesthetic appearance of the umbilicus).
  Patient's level of importance regarding the aesthetic appearance of the umbilicus was recorded preoperatively (right before the surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie McFadden, M.D, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No